CLINICAL TRIAL: NCT01716117
Title: The Surpass Intracranial Aneurysm Embolization System Pivotal Trial to Treat Large or Giant Wide Neck Aneurysms (SCENT Trial)
Brief Title: Safety and Effectiveness of an Intracranial Aneurysm Embolization System for Treating Large or Giant Wide Neck Aneurysms
Acronym: SCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-04
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Brain Aneurysm
Keywords: Large aneurysm; Giant aneurysm; Wide neck aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: The SCENT Trial is a multi-center, prospective, non-randomized trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surpass Flow Diverter (Experimental): The objective of this study is to determine the safety and effectiveness of the Surpass Flow Diverter (Surpass System) in the endovascular treatment of large or giant wide-necked intracranial aneurysms in the internal carotid artery up to the terminus.
  Interventions: Device: Surpass Flow Diverter

INTERVENTIONS:
Device: Surpass Flow Diverter — Treatment of an intracranial aneurysm involves the placement of a specially designed metallic mesh tube in a vessel in the brain where an aneurysm is located. The device looks like a fishnet sock with both ends open. Each device is delivered through a small catheter (a long, flexible tube). The catheter containing the device is inserted and advanced into a vessel in the brain. The device is then placed in the brain vessel by releasing it from the catheter. Once the device is placed inside the brain vessel, it is intended to reinforce the area of the vessel that is weakened and bulging (the aneurysm), and to cause blood to flow down the vessel and away from the aneurysm while allowing blood in the aneurysm to clot. This procedure is called an endovascular aneurysm treatment because the device is delivered through the blood vessels.
  Other Names: Flow diverter; Endovascular aneurysm treatment

SUMMARY:
This clinical research study is designed to determine safety and effectiveness of the Surpass Flow Diverter (Surpass System), an investigational device developed to treat wide-neck, large or giant intracranial aneurysms. An intracranial aneurysm is a bulge in the wall of a blood vessel in the brain. The bulge is caused by a weakening of the vessel wall. If left untreated, the bulge may continue to grow larger and ultimately the vessel may break open (rupture), resulting in serious bleeding into or around the brain. The information collected from this study will be used to evaluate how well patients do when treated with the Surpass System both immediately after treatment of an aneurysm and over a long period of time (5 years).

DETAILED DESCRIPTION:
The objective of this study is to determine safety and effectiveness of the Surpass Flow Diverter (Surpass System) in the endovascular treatment of large or giant wide-necked intracranial aneurysms in the internal carotid artery up to the terminus. The Surpass Flow Diverter is an intracranial implant designed to be placed in a parent artery so as to divert blood flow away from an aneurysm. Use of the Surpass System may be associated with a decrease in neurological death or ipsilateral stroke in patients with large or giant wide-neck aneurysms. In a given patient, the Surpass System will be deemed effective if treatment results in complete occlusion of their aneurysm without clinically significant stenosis of the parent artery, or requires retreatment of the aneurysm through 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 80 years
* Subject or legal representative is willing and able to give informed consent
* Subject has a single targeted intracranial aneurysm
* Subject agrees to return to the treating Investigator for all scheduled follow up visits and is capable of returning to the hospital for follow up

Exclusion Criteria:

* Known allergy or contraindication to aspirin, clopidogrel/Plavix, heparin, local or general anesthesia
* Known history of life threatening allergy to contrast dye
* Known allergy to nickel, chromium cobalt, tungsten or platinum
* Subject has documented resistance to clopidogrel/Plavix
* Major surgery within previous 30 days or planned in the next 120 days after enrollment date
* Previous intracranial implant associated with the symptomatic distribution within the past 12 weeks prior to treatment date
* Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to treatment date
* Any previous stenting of parent artery at or proximal to the aneurysm where it would interfere with the placement and proper apposition of the device
* Any previous coiling where it would interfere with the placement and proper apposition of the device
* Platelet count less than 100,000 cells/mm3 or known platelet dysfunction
* More than one intracranial aneurysm (IA) that requires treatment within 12 months
* Asymptomatic extradural aneurysms requiring treatment
* Contraindication to CT scan or MRI
* Severe neurological deficit that renders the subject incapable of living independently
* Unstable neurological deficit (i.e., worsening of clinical condition in the last 30 days)
* Evidence of active infection at the time of treatment
* Dementia or psychiatric problem that prevents the patient from completing required follow up
* Co-morbid conditions that may limit survival to less than 24 months
* Serum creatinine greater or equal to 2.5 mg/dL
* Female subjects who are pregnant or planning to become pregnant within the study period
* Subject with anatomy not appropriate for endovascular treatment due to severe intracranial vessel tortuosity or stenosis
* Extra-cranial stenosis or parent vessel with stenosis greater than 50% in the area proximal to the aneurysm
* Other known serious concurrent medical conditions
* History of intracranial vasospasm not responsive to medical therapy
* Subject with an intracranial mass, or is undergoing radiation therapy for carcinoma or sarcoma of the head or neck region
* Subject has a history of bleeding diathesis or coagulopathy, international normalized ratio (INR) greater than 1.5, or will refuse blood transfusions
* Subject had a subarachnoid hemorrhage within 30 days prior to the enrollment date
* Subject has a non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm
* Inability to understand the study or a history of non-compliance with medical advice
* Current use of illicit substance
* Enrollment in another trial involving an investigational product
* Subject has a need for long-term use of anticoagulants (i.e., Warfarin, Dabigatran)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-10-25 (Actual); Primary Completion 2016-12-11 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Hanel, MD, PhD, Principal Investigator — Lyerly Baptist Medical Center, Jacksonville, Florida; Philip M Meyers, MD, Principal Investigator — Columbia University
Locations (26):
- United States (25):
  - University of California, Irvine, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - University of Florida, Gainesville, Florida
  - Lyerly Neurosurgery/Baptist Health System, Jacksonville, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - University at Buffalo, Buffalo, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Fort Sanders Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas - Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- UMC St Radboud, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD information available to other researchers. Blinded study data by mITT and Roll-in cohorts may be made available to SCENT researchers post publication of the primary study results.

REFERENCES:
- [Derived] Meyers PM, Coon AL, Kan P, Dogan A, Bain M, Welch BG, Ebersole K, De Vries J, Wakhloo AK, Taussky P, Jenkins P, Hanel RA; SCENT Investigators. Five-year results of the SCENT trial with Surpass flow diverters to treat large or giant wide-neck aneurysms. J Neurointerv Surg. 2025 Sep 12;17(10):1078-1082. doi: 10.1136/jnis-2024-022977. PMID 40335285
- [Derived] Hanel RA, Cortez GM, Coon AL, Kan P, Taussky P, Wakhloo AK, Welch BG, Dogan A, Bain M, De Vries J, Ebersole K, Meyers PM; SCENT Investigator Group. Surpass Intracranial Aneurysm Embolization System Pivotal Trial to Treat Large or Giant Wide-Neck Aneurysms - SCENT: 3-year outcomes. J Neurointerv Surg. 2023 Nov;15(11):1084-1089. doi: 10.1136/jnis-2022-019512. Epub 2022 Nov 14. PMID 36375835
- [Derived] Kan P, Mohanty A, Meyers PM, Coon AL, Wakhloo AK, Marosfoi M, Bain M, de Vries J, Ebersole K, Lanzino G, Taussky P, Hanel RA. Treatment of large and giant posterior communicating artery aneurysms with the Surpass streamline flow diverter: results from the SCENT trial. J Neurointerv Surg. 2023 Jul;15(7):679-683. doi: 10.1136/neurintsurg-2021-018189. Epub 2022 May 12. PMID 35551072
- [Derived] Meyers PM, Coon AL, Kan PT, Wakhloo AK, Hanel RA. SCENT Trial. Stroke. 2019 Jun;50(6):1473-1479. doi: 10.1161/STROKEAHA.118.024135. Epub 2019 May 14. PMID 31084335
- [Derived] Colby GP, Lin LM, Caplan JM, Jiang B, Michniewicz B, Huang J, Tamargo RJ, Coon AL. Flow diversion of large internal carotid artery aneurysms with the surpass device: impressions and technical nuance from the initial North American experience. J Neurointerv Surg. 2016 Mar;8(3):279-86. doi: 10.1136/neurintsurg-2015-011769. Epub 2015 May 18. PMID 25987590

RESULTS

PARTICIPANT FLOW:
Groups:
- Surpass Flow Diverter (mITT Population): The mITT population was defined in the clinical protocol as all enrolled subjects for whom the investigational device entered the body, regardless of whether or not the device was successfully implanted.
- Surpass Flow Diverter (Roll-In Population): An additional 45 "Roll-In" subjects were permitted in the original approved clinical protocol, which was updated to allow for up to 70 "Roll-In" and "Enrolled but Not Treated" subjects. Data from this population were not included in the mITT Primary Endpoint analysis. Neither did they serve as a control population. Results are displayed for informational purposes.
Period: Overall Study
Arm/Group | Surpass Flow Diverter (mITT Population) | Surpass Flow Diverter (Roll-In Population)
Started | 180 | 33
Discharge | 177 | 33
1-Month Visit | 176 | 33
6-Month Visit | 174 | 32
Completed | 173 | 31
Not Completed | 7 | 2
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surpass Flow Diverter (mITT): The mITT population was defined in the clinical protocol as all enrolled subjects for whom the investigational device entered the body, regardless of whether or not the device was successfully implanted.
- Roll-In: An additional 45 "Roll-In" subjects were permitted in the original approved clinical protocol, which was updated to allow for up to 70 "Roll-In" and "Enrolled but Not Treated" subjects. Data from this population were not included in the mITT Primary Endpoint analysis. Neither did they serve as a control population. Results are displayed for informational purposes.
- Total: Total of all reporting groups
Arm/Group | Surpass Flow Diverter (mITT) | Roll-In | Total
Number analyzed (Participants) | 180 | 33 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.9) | 62.4 (11.1) | 61.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 29 | 194
  Male | 15 | 4 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects may contribute toward more than one criterion for race. The total count may exceed the number of study subjects in each study cohort.
  Participants
    American Indian/Alaska Native | 2 | 0 | 2
    Asian | 6 | 2 | 8
    Black or African American | 26 | 7 | 33
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    White | 140 | 22 | 162
    Other | 2 | 2 | 4
    Not Reported | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 4 | 18
  Not Hispanic or Latino | 158 | 29 | 187
  Unknown | 6 | 0 | 6
  Not Reported | 2 | 0 | 2
Age [Median (Inter-Quartile Range); unit: years] | 61.5 [38.0 to 80.0] | 65.0 [39.0 to 79.0] | 62.0 [38.0 to 80.0]
Height [Mean (Standard Deviation); unit: inches (in)] | 64.8 (3.2) | 64.3 (3.6) | 64.7 (3.3)
Height [Median (Inter-Quartile Range); unit: inches (in)] | 65.0 [52.0 to 75.0] | 64.2 [59.1 to 72.0] | 65.0 [52.0 to 75.0]
Weight [Mean (Standard Deviation); unit: pounds (lbs)] | 166.0 (40.2) | 154.5 (31.6) | 164.2 (39.1)
Weight [Median (Inter-Quartile Range); unit: pounds (lbs)] | 158.4 [83.6 to 281.6] | 149.6 [95.0 to 215.6] | 158.4 [83.6 to 281.6]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: lbs/in^2] | 27.8 (6.1) | 26.3 (4.5) | 27.5 (5.9)
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: lbs/in^2] | 27.0 [16.0 to 49.0] | 26.0 [18.0 to 35.0] | 27.0 [16.0 to 49.0]
Smoking Status/Alcohol Use [Count of Participants; unit: Participants] — Subjects may contribute toward more than one criterion for smoking status.
  Participants
    Current Smoker | 36 | 10 | 46
    Past Smoker | 79 | 11 | 90
    Current Consumer of Alcohol | 91 | 12 | 103

OUTCOME MEASURES:

1. Primary Outcome: mITT Primary Effectiveness Endpoint. Based on Subjects With 100% Occlusion of the Aneurysm Without Clinically Significant Stenosis of the Parent Artery, and Without Any Subsequent Treatment of the Target Aneurysm at the 12 Month Follow up Visit.
Description: Percent of subjects with 100% occlusion of the aneurysm without clinically significant stenosis (defined as less than or equal to 50% stenosis) of the parent artery based on core lab evaluation of the 12 month follow up angiogram and without any subsequent treatment of the target aneurysm at the 12 month follow up visit.
Time Frame: 12 months
Population: The mITT primary endpoint analysis population (n = 180) is based on subjects in the mITT arm and does not include the results of subjects treated in the Roll-in population (n = 33).
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Surpass Flow Diverter (mITT Population)
Number analyzed (Participants) | 180
Percent of participants
  Primary Effectiveness Endpoint Composite Success | 62.8 [55.3 to 69.9]
  Parent Artery Stenosis > 50% | 3.3 [1.2 to 7.1]
  Retreatment of Target Intracranial Aneurysm | 0.6 [0.0 to 3.1]

2. Primary Outcome: mITT Primary Safety Endpoint. Based on Subjects Experiencing Neurologic Death or Major Ipsilateral Stroke Through 12 Month Follow-up.
Description: Subjects experiencing neurologic death or major ipsilateral stroke through 12 months.
Time Frame: 12 months
Population: The mITT primary endpoint analysis population (n = 180) is based on subjects in the mITT arm and does not include the results of subjects treated in the Roll-in arm (n = 33).
Measure: Count of Participants; unit: Participants
Arm/Group | Surpass Flow Diverter (mITT)
Number analyzed (Participants) | 180
Participants
  Major Ipsilateral Stroke | 19
  Neurological Death | 5
  Primary Safety Endpoint Failure | 19

3. Secondary Outcome: Raymond-Roy Score Per Core Lab Assessment Based on Device Apposition at 12 Months Post-Procedure
Description: The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete obliteration (best); Class II: residual neck; Class III: residual aneurysm (worse).
Time Frame: 12 months
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Device Not Fully Apposed to Vessel Wall at 12 Months: Subgroups of patients who did not have full apposition of the device to the vessel wall.
- Device Fully Apposed to Vessel Wall at 12 Months: Subgroups of patients who had full apposition of the device to the vessel wall.
Arm/Group | Device Not Fully Apposed to Vessel Wall at 12 Months | Device Fully Apposed to Vessel Wall at 12 Months
Number analyzed (Participants) | 34 | 125
Participants
  Raymond-Roy I | 17 | 99
  Raymond-Roy II | 3 | 14
  Raymond-Roy III | 14 | 12

4. Other Pre Specified Outcome: Clinical Events Committee (CEC) Adjudicated Rate of Minor Strokes Through 12 Month Follow-Up
Description: Patients with minor strokes through 12 months
Time Frame: 12 Months
Population: Secondary endpoint analysis of the mITT population (n = 180) are presented herein for comparison to results of subjects in the Roll-in population (n = 33).
Measure: Count of Participants; unit: Participants
Arm/Group | Surpass Flow Diverter (mITT Population) | Surpass Flow Diverter (Roll-In Population)
Number analyzed (Participants) | 180 | 33
Participants | 12 | 1

5. Other Pre Specified Outcome: Subgroup Analysis of Primary Effectiveness Endpoint Based on Subject Age ≥ 65 Years Versus < 65 Years in mITT Population
Description: Primary effectiveness by age group
Time Frame: 12 Months
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Under Age 65: Subjects below 65 years of age
- Age 65 and Older: Subjects of at least 65 years of age
Arm/Group | Under Age 65 | Age 65 and Older
Number analyzed (Participants) | 114 | 66
Participants | 80 | 33

6. Other Pre Specified Outcome: CEC Adjudicated Primary Effectiveness Endpoint Outcomes for Giant and Non-Giant (Large) Intracranial Aneurysms Through 12 Month Follow-Up - mITT Population
Description: Primary effectiveness by intracranial aneurysm size
Time Frame: 12 Months
Population: mITT Population
Measure: Count of Participants; unit: Participants
Groups:
- All Intracranial Aneurysm Sizes Except Giant: Intracranial aneurysms not considered giant
- Giant Intracranial Aneurysms: Intracranial aneurysms considered giant
Arm/Group | All Intracranial Aneurysm Sizes Except Giant | Giant Intracranial Aneurysms
Number analyzed (Participants) | 167 | 13
Participants | 107 | 6

7. Other Pre Specified Outcome: Number of Surpass Streamline Flow Diverters Implanted Per Subject in SCENT Trial - mITT and Roll-In Populations
Description: Number of devices implanted in subjects by study population
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- Roll-In: An additional 45 "Roll-In" subjects were permitted in the original approved clinical protocol, which was updated to allow for up to 70 "Roll-In" and "Enrolled but Not Treated" subjects.
Arm/Group | Surpass Flow Diverter (mITT) | Roll-In
Number analyzed (Participants) | 180 | 33
Participants
  None | 3 | 0
  One | 156 | 25
  Two | 21 | 7
  >2 | 0 | 1

8. Post Hoc Outcome: Post-Hoc Primary Safety Endpoint of Disabling Stroke or Neurologic Death Through 12 Month Follow-Up
Description: Subjects experiencing neurologic death or disabling stroke through 12 months.
Time Frame: 12 Months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Surpass Flow Diverter (mITT)
Number analyzed (Participants) | 180
Percent of participants
  Disabling Stroke or Neurologic Death | 6.1 [3.1 to 10.7]
  Neurologic Death | 2.8 [0.9 to 6.4]
  Disabling Stroke | 6.1 [3.1 to 10.7]

ADVERSE EVENTS:
Time Frame: Through 12 Months Post Procedure
Description: The definition of adverse event and/or serious adverse event used during the collection of adverse event information was consistent with that listed above in the clinicaltrials.gov definitions. Adverse events and serious adverse events were organized by System/Organ Class and Preferred Term.
Groups:
- Surpass Flow Diverter (Roll-in Population): The Roll-in population was defined in the clinical protocol as all subjects who were enrolled as training cases and not considered part of the mITT population, and in whom the Surpass™ Flow Diverter entered the body regardless of whether or not the device was successfully implanted.
Arm/Group | Surpass Flow Diverter (mITT Population) | Surpass Flow Diverter (Roll-in Population)
All-Cause Mortality (participants affected / at risk) | 5/180 | 2/33
Serious Adverse Events (participants affected / at risk) | 54/180 | 17/33
Other Adverse Events (participants affected / at risk) | 129/180 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surpass Flow Diverter (mITT Population) (N=180) | Surpass Flow Diverter (Roll-in Population) (N=33)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 1 (1)
Retinal Infarction (Eye disorders) | 2 (2) | 0 (0)
Visual Impairment (Eye disorders) | 2 (2) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal Hematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 3 (3) | 0 (0)
Thrombosis in Device (General disorders) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Vascular Pseudo-Aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhagic Stroke (Nervous system disorders) | 4 (4) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Ischemic Stroke (Nervous system disorders) | 11 (11) | 3 (3)
Subarachnoid Hemorrhage (Nervous system disorders) | 5 (5) | 2 (2)
Syncope (Nervous system disorders) | 4 (4) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 3 (3) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Intra-Cerebral Aneurysm Operation (Surgical and medical procedures) | 3 (3) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Anginia Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Optic Ischaemic Neuropathy (Eye disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Pseudocyst (General disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Optic Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
VIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aneurysm Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arterial Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombotic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral Salt-Wasting Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mental Status Changes Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device Occlusion (General disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surpass Flow Diverter (mITT Population) (N=180) | Surpass Flow Diverter (Roll-in Population) (N=33)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Visual Impairment (Eye disorders) | 14 (14) | 4 (4)
Diplopia (Eye disorders) | 7 (7) | 0 (0)
Eye Pain (Eye disorders) | 8 (8) | 0 (0)
Vision Blurred (Eye disorders) | 7 (7) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Dry Eye (Eye disorders) | 2 (2) | 0 (0)
Eye Pruritis (Eye disorders) | 2 (2) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal Hemorrhage (Eye disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mouth Hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal Hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal Hematoma (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 10 (10) | 0 (0)
Thrombosis in Device (General disorders) | 2 (2) | 0 (0)
Catheter Site Hemorrhage (General disorders) | 4 (4) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 4 (4) | 0 (0)
Gait Disturbance (General disorders) | 3 (3) | 0 (0)
Implant Site Pain (General disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 10 (10) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 9 (9) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular Pseudo-Aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neurological Examination Abnormal (Investigations) | 4 (4) | 0 (0)
Carotid Bruit (Investigations) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 12 (12) | 0 (0)
Reversible Ischemic Neurological Deficit (Nervous system disorders) | 12 (12) | 0 (0)
Hypoesthesia (Nervous system disorders) | 7 (7) | 2 (2)
Transient Ischemic Attack (Nervous system disorders) | 3 (3) | 0 (0)
Amnesia (Nervous system disorders) | 3 (3) | 0 (0)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 4 (4) | 0 (0)
Migraine (Nervous system disorders) | 4 (4) | 0 (0)
Aphasia (Nervous system disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Third Nerve Paralysis (Nervous system disorders) | 2 (2) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Restless Leg Syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Confusional State (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 10 (10) | 2 (2)
Hematoma (Vascular disorders) | 7 (7) | 0 (0)
Vasospasm (Vascular disorders) | 6 (6) | 0 (0)
Hemorrhage (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Orithostatic Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Vitreous Floaters (Eye disorders) | 3 (3) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 52 (52) | 14 (14)
Pupils Unequal (Eye disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research parties agree not to make any publication of study results, including without limitation the study data, until completion of the study and publication of the multi-center results in a peer-reviewed journal. Thereafter, the research parties may publish their individual site experience.